CLINICAL TRIAL: NCT02160067
Title: A Four-period, Randomised, Open-label, Crossover, Pharmacokinetic Study to Assess the Dose Proportionality and Relative Bioavailability of Buprenorphine Transdermal Delivery System Second Generation Patches Compared to First Generation Patches, in Healthy Volunteers
Brief Title: A Dose Proportionality and Bioavailability Assessment of Buprenorphine Transdermal Delivery System Second Generation Patches
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BUP1506; 2014-000691-26 (EudraCT Number)
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Healthy Volunteers; Pharmacokinetics
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Second generation patch BTDS 12.6mg
  Interventions: Drug: Second generation BTDS patch
- Treatment B (Experimental): Second generation patch BTDS 3.15mg
  Interventions: Drug: Second generation BTDS patch
- Treatment C (Active Comparator): First generation patch BuTrans 20mg
  Interventions: Drug: First generation BuTrans patch
- Treatment D (Active Comparator): First generation patch BuTrans 5mg
  Interventions: Drug: First generation BuTrans patch

INTERVENTIONS:
Drug: Second generation BTDS patch
  Arms: Treatment A; Treatment B
Drug: First generation BuTrans patch
  Arms: Treatment C; Treatment D

SUMMARY:
The purpose of this study is to obtain pharmacokinetic data for a dose proportionality and relative bioavailability assessment of 2nd generation BTDS patches compared to 1st generation BTDS patches.

DETAILED DESCRIPTION:
The objective is to examine a new 2nd generation BTDS patch formulation at 2 strengths: 3.15 mg and 12.6 mg, compared to 1st generation patches at 2 strengths: 5 mg and 20 mg, to assess dose proportionality and relative bioavailability before proceeding to a definitive program of studies. Determination is by measurement of drug concentrations in the blood at serial collection time points pre-dose until 288 hours post-patch application.

ELIGIBILITY:
Inclusion Criteria

1. Provide written informed consent.
2. Healthy male or female subjects aged 18 to 55 inclusive.
3. Female subjects of child bearing potential must be willing to use two highly effective methods of contraception throughout the study, one of which must include a barrier method. .
4. Male subjects who are willing to use contraception with their partners throughout the study and for 30 days after completion of the study and agree to inform the Investigator if their partner becomes pregnant during this time.
5. Body weight ranging from 55 to 100 kg and a BMI ≥ 18.5 and ≤ 29.9.
6. Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
7. Willing to eat all the food supplied throughout the study.
8. The subject's primary care physician has confirmed within the last 12 months that there is nothing in the subject's medical history that would preclude their enrolment into a clinical study.
9. Will refrain from strenuous exercise during the entire study.

Exclusion criteria

1. Female subjects who are pregnant or lactating.
2. Any history of drug or alcohol abuse.
3. Any history of conditions that might interfere with drug absorption, distribution, metabolism or excretion.
4. Use of opioid or opioid antagonist-containing medication in the past 30 days.
5. Any history of frequent nausea or vomiting regardless of aetiology.
6. Any history of seizures or symptomatic head trauma.
7. Participation in a clinical drug study during the 90 days preceding the initial dose in this study, participation in the previous Mundipharma Research Ltd, BUP1505 study or participation in any other study during this study.
8. Any significant illness during the 4 weeks preceding entry into this study.
9. A history of additional risk factors for Torsades de Pointes (e.g. heart failure, hypokalaemia, personal or family history of long QT syndrome, syncope, or family history of sudden death).
10. Abnormal cardiac conditions including any of the following:
11. Use of medication within 5 times the half-life or minimum 14 days for prescription medication or 7 days for over-the-counter preparations (including vitamins, herbal and/or mineral supplements), whichever is longer, before the first dose of study treatment and during the study (with the exception of the continued use of HRT and contraceptives).
12. Refusal to abstain from caffeine or xanthine containing beverages and grapefruit juice within 48 hours before IMP administration until after the last study PK sample has been taken in each study period.
13. Weekly alcohol intake exceeding the equivalent of 14 units/week for females and 21 units/week for males.
14. Consumption of alcoholic beverages within 48 hours before IMP administration, and refusal to abstain from alcohol for the duration of the study confinement and for at least 48 hours after the last naltrexone dose in each study period.
15. History of smoking within 45 days of IMP administration and refusal to abstain from smoking during the study.
16. Blood or blood products donated within 90 days prior to IMP administration or any time during the study, except as required by this protocol.
17. Positive results of urine drug screen, alcohol test, pregnancy test, HBsAg, Hepatitis C antibody, or HIV tests.
18. Known sensitivity to buprenorphine, naltrexone, related compounds or any of the excipients or any contraindications as detailed in the Butrans Summary of Product Characteristics or Nalorex Summary of Product Characteristics.
19. Clinically significant history of allergic reaction to wound dressings or elastoplast.
20. Subjects with any dermatological disorder or tattoos at the proposed sites of patch application, or with a history of eczema/cutaneous atrophy.
21. Subjects who will not allow hair to be removed at the proposed patch application sites which may prevent proper placement of the patch.
22. Refusal to allow their primary care physician to be informed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters | Up to 288 hours
  AUC and Cmax

SECONDARY OUTCOMES:
Adverse events | 7 to 10 days
  AEs will be recorded through spontaneous reporting

OTHER OUTCOMES:
Vital Signs composite measure | 0-288 hours
  Vital signs are collected as a composite measure- blood pressure, pulse rate, tympanic temperature, respiration rate, SpO2
Clinical Laboratory Tests | Day 0 and Day 7-10
  Blood samples will be taken at screening, pre dose, 192 hours, and post study medical for routine blood chemistry and urinalysis
ECG | Screening, pre dose, 72, 120, 168hours, and day 7-10
  ECGs

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical Ltd, Nottingham, United Kingdom